CLINICAL TRIAL: NCT00168025
Title: A Multicenter Study on the Efficacy, Safety and Pharmacokinetics of IgPro10 in Patients With Primary Immunodeficiency (PID)
Brief Title: Efficacy and Safety of Intravenous Immunoglobulin IgPro10 in Patients With Primary Immunodeficiencies (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB03_002CR
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency
Keywords: Immunoglobulin Intravenous; Agammaglobulinemia; Hypogammaglobulinemia; Common variable immunodeficiency; Immunoglobulin G; Children
MeSH Terms: conditions — Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency | interventions — Immunoglobulins, Intravenous

ARMS (1):
- IgPro10 (Experimental)
  Interventions: Drug: Immunoglobulins Intravenous (Human)

INTERVENTIONS:
Drug: Immunoglobulins Intravenous (Human)

SUMMARY:
The purpose of this study is to demonstrate the effect of IgPro10 on the prevention of serious bacterial infections in patients with primary immunodeficiency.

As secondary endpoints the rate of overall infections, the tolerability and safety of IgPro10 are studied.

A part of the patients are participating in a pharmacokinetic substudy.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with primary immunodeficiency
* Patients who have received stable IVIG therapy at 3- or 4-weekly intervals for at least 6 months

Key Exclusion Criteria:

* Newly diagnosed PID
* Allergic reactions to immunoglobulins or other blood products
* Administration of steroids (daily ≥ 0.15 mg prednisone equivalent/kg/day) or other immunosuppressive drugs
* Concomitant diseases such as hypoalbuminemia, protein-losing enteropathies, kidney diseases with proteinuria, malignancies of lymphoid cells (e.g. lymphocytic leukemia), and recent history of migraine
* History of cardiac insufficiency (NYHA III/IV), cardiomyopathy, congestive heart failure, severe hypertension

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-09; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Annualized rate of acute serious bacterial infections

SECONDARY OUTCOMES:
Number of infections
Number of days out of work / school due to underlying PID
Adverse events temporally associated with study drug infusion
Trough levels of total IgG serum concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring

REFERENCES:
- [Background] Sleasman JW, Duff CM, Dunaway T, Rojavin MA, Stein MR. Tolerability of a new 10% liquid immunoglobulin for intravenous use, Privigen, at different infusion rates. J Clin Immunol. 2010 May;30(3):442-8. doi: 10.1007/s10875-010-9373-x. Epub 2010 Mar 10. PMID 20217199
- [Result] Stein MR, Nelson RP, Church JA, Wasserman RL, Borte M, Vermylen C, Bichler J; IgPro10 in PID study group. Safety and efficacy of Privigen, a novel 10% liquid immunoglobulin preparation for intravenous use, in patients with primary immunodeficiencies. J Clin Immunol. 2009 Jan;29(1):137-44. doi: 10.1007/s10875-008-9231-2. Epub 2008 Sep 24. PMID 18814020